CLINICAL TRIAL: NCT07392515
Title: Cognitive and Motor Recovery in Frail Patients With Hip Fracture: Effectiveness of Digital Technology-Assisted Rehabilitation and Analysis of Biomolecular Mechanisms
Brief Title: Cognitive and Physical Recovery After Hip Fracture in Frail Patients Using Digital Rehabilitation Technology
Acronym: FEWF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.T. Cure Ortopediche Traumatologiche S.p.A. (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Ennio Ferlazzo, Head of Rehabilitation Department, C.O.T. Cure Ortopediche Traumatologiche S.p.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNC0000007-B53C22006770008
Record Dates: First submitted 2026-01-13; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Fracture Femur; Hip Arthroplasty Replacement; Total Hip Arthroplasty (THA)
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation (Active Comparator): Patients receive a standard inpatient conventional rehabilitation program including joint mobilization, postural re-education, muscle strengthening, and gait training with assistive devices.
  Interventions: Other: Conventional rehabilitation intervention
- Technology-Assisted Integrated Rehabilitation (Experimental): Patients receive an integrated rehabilitation program combining sensor-based technology-assisted training (1/3 of daily sessions) with conventional rehabilitation (2/3 of daily sessions).
  Interventions: Device: Experimental intervention - integrated treatment with a sensor-based device

INTERVENTIONS:
Device: Experimental intervention - integrated treatment with a sensor-based device — The technology/robotic group will perform one-third (1/3) of the daily rehabilitation using technology-assisted devices and two-thirds (2/3) using conventional rehabilitation. In addition to the conventional rehabilitation described below, the treatment will include technology-assisted rehabilitation consisting of facilitated active joint mobilization exercises with visual and auditory feedback, aimed at stimulating motor and cognitive functions, as well as gait training.
  Arms: Technology-Assisted Integrated Rehabilitation
Other: Conventional rehabilitation intervention — The conventional rehabilitation programme includes assisted and facilitated joint mobilization exercises to improve range of motion; exercises for postural readaptation of the trunk to the upright position; isometric exercises; and gait training using a 4-wheeled walker or forearm crutches (Canadian crutches), aimed at improving walking ability and achieving an appropriate recovery of the gait pattern.
  Arms: Conventional Rehabilitation

SUMMARY:
The aim of this study is to evaluate whether integrating a technology-based rehabilitation approach with conventional therapies in the rehabilitation of patients with proximal femoral fracture may be advantageous compared with conventional therapy alone. Specifically, the objective is to assess whether the addition of technology-assisted rehabilitation can improve cognitive function, in addition to motor function and overall abilities, compared with conventional rehabilitation alone. Furthermore, the study intends to explore the feasibility of implementing technology-assisted rehabilitation as a stable and routine component of everyday clinical practice, also considering the perspective of healthcare professionals.

DETAILED DESCRIPTION:
This is a national, multicenter, non-profit, post-market interventional longitudinal clinical study designed to evaluate the effectiveness of integrating technology-assisted rehabilitation with conventional rehabilitation in elderly patients undergoing inpatient rehabilitation after surgically treated proximal femoral fracture.

Eligible participants aged 65 to 89 years who have undergone surgical treatment for proximal femoral fracture (total hip arthroplasty, partial hip arthroplasty, or intramedullary nailing) and who are clinically stable will be enrolled during their inpatient rehabilitation stay. After enrollment, patients will be randomly assigned to one of two treatment arms: (1) conventional rehabilitation alone (control group) or (2) integrated rehabilitation combining conventional therapy with sensor-based technology-assisted rehabilitation (experimental group). Randomization will be centralized and stratified by center and age group.

The total rehabilitation program consists of 18 sessions delivered over approximately 3-4 weeks, with a frequency of 5-6 sessions per week. Patients in the experimental group will perform approximately one-third of daily rehabilitation sessions using sensor-based digital devices providing real-time visual and auditory feedback, and two-thirds with conventional rehabilitation. Technology-assisted training includes facilitated active joint mobilization, motor and cognitive stimulation tasks, and gait training. The control group will receive conventional rehabilitation only, including assisted joint mobilization, postural re-education, muscle strengthening exercises, and gait training with assistive devices.

Clinical assessments will be performed at baseline (T0) and at the end of the rehabilitation program (T1). Motor performance will be assessed using the Timed Up and Go (TUG) test, which measures the time required for a participant to stand up from a chair, walk three meters, turn around, walk back, and sit down, as well as the Timed Up and Go Dual Task (TUG Dual Task), which evaluates mobility under simultaneous cognitive or motor task conditions. Additional functional outcomes include the Harris Hip Score, Barthel Index, pain assessed by Numeric Rating Scale, and health-related quality of life assessed by the SF-36. Cognitive status will be assessed using the Mini-Mental State Examination (MMSE). Blood samples will be collected at T0 and T1 to measure serum brain-derived neurotrophic factor (BDNF) levels and to analyze the rs6265 (Val66Met) polymorphism.

The primary endpoints are the change in serum BDNF levels and the change in TUG and TUG Dual Task performance from baseline to the end of treatment. Secondary endpoints include changes in functional scores, pain, quality of life, and exploratory analysis of the BDNF genetic polymorphism.

Healthcare professionals involved in the rehabilitation program will also complete the Work-Related Quality of Life (WRQoL) questionnaire to explore the perceived impact of technology-assisted rehabilitation on work-related quality of life.

Statistical analysis will be performed to evaluate differences between the control and experimental groups and changes over time in outcome measures. A p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 89 years
* Patients who have undergone one of the following surgical treatments specifically for proximal femur fracture including Total hip arthroplasty (total hip replacement), Partial hip arthroplasty (hemiarthroplasty), Intramedullary nailing
* Time since surgery not exceeding 15 days
* Clinical stability
* Patients admitted to the rehabilitation wards of the centers involved in the study and therefore eligible for rehabilitative therapy.

Exclusion Criteria:

* Age > 90 years
* Age < 65 years
* Refusal to sign the informed consent form
* Behavioral or cognitive disorders limiting compliance with the rehabilitative treatment
* Presence of mechanical instability of the implanted surgical device
* Clinical instability (e.g., sepsis, severe anemia, cardiorespiratory failure) or pre-existing comorbidities affecting ambulation (neurological diseases or chronic pre-existing disabilities)
* Concomitant presence of other fractures that prevent the possibility of carrying out a rehabilitative treatment
* Severe visual impairments not correctable with lenses that prevent the patient from performing the treatment using digital tools
* Pre-existing motor disability prior to the femur fracture due to other systemic diseases (e.g., advanced-stage neurodegenerative diseases, severe heart failure)
* Conditions contraindicating the use of sensors (pacemaker, epilepsy, skin lesions, open wounds, and severe allergies in areas of contact with the devices).

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in serum BDNF levels | Baseline and within 3 days after completion of the rehabilitative treatment
  Difference in serum brain-derived neurotrophic factor (BDNF) levels between baseline and the end of the rehabilitative treatment, assessed to evaluate biomolecular changes associated with neuroplasticity.
Change in Timed Up and Go test | Baseline and within 3 days after completion of the rehabilitative treatment
  Difference in functional mobility, balance, and gait performance assessed using the Timed Up and Go test between baseline and end of rehabilitative treatment.
Change in Timed Up and Go Dual Task test | Baseline and within 3 days after completion of the rehabilitative treatment
  Difference in cognitive-motor dual-task performance assessed using the Timed Up and Go Dual Task test between baseline and end of rehabilitative treatment.

SECONDARY OUTCOMES:
Change in the Harris Hip Score (HHS) | Baseline and within 3 days after completion of the rehabilitative treatment
  Change in hip function, pain, and functional ability as assessed by the Harris Hip Score, a clinician-administered outcome measure ranging from 0 to 100 points, where higher scores indicate better hip function, assessed at baseline and at the end of the rehabilitative treatment.
Change in the modified Barthel Index | Baseline and within 3 days after completion of the rehabilitative treatment
  Change in independence in activities of daily living as assessed by item-level scores of the Barthel Index, a validated measure of functional independence ranging from 0 to 100 points, where higher scores indicate greater independence, assessed at baseline and at the end of the rehabilitative treatment (Italian version, 2015).
Change in pain intensity measured by the Numeric Rating Scale (NRS) | Baseline and within 3 days after completion of the rehabilitative treatment
  Change in pain intensity as assessed by the Numeric Rating Scale, a patient-reported outcome measure ranging from 0 to 10, where higher scores indicate greater pain intensity, assessed at baseline and at the end of the rehabilitative treatment.
Change in quality of life measured by the SF-36 | Baseline and within 3 days after completion of the rehabilitative treatment
  Change in health-related quality of life as assessed by the 36-Item Short Form Health Survey (SF-36), a validated patient-reported outcome measure composed of multiple domains, each scored on a 0 to 100 scale, where higher scores indicate better health-related quality of life, assessed at baseline and at the end of the rehabilitative treatment.
Analysis of the rs6265 polymorphism (Val66Met mutation) of the BDNF gen | Baseline
  Genotyping of the BDNF rs6265 (Val66Met; G196A) single-nucleotide polymorphism to classify participants as Val/Val, Val/Met, or Met/Met and explore its association with serum BDNF levels and rehabilitative outcomes.
Healthcare professionals' perspective on work-related quality of work in the two different treatment approaches. | At the end of treatment delivery for both interventions
  Assessment of healthcare professionals' work-related quality of life using the Work-Related Quality of Life Scale (WRQoL).
  The WRQoL total score ranges from 23 to 115, with higher scores indicating better perceived work-related quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - COT - Cure Ortopediche Traumatologiche, Messina, Italy
  - Fondazione Don Carlo Gnocchi - Centro Santa Maria della Provvidenza, Roma, Italy

IPD SHARING:
Plan to Share IPD: No